CLINICAL TRIAL: NCT01201057
Title: A Double-blind, Multi-center, Randomized, Placebo Controlled, Dose-ranging Study to Determine the Efficacy and Safety of SPL7013 Gel (VivaGel®) Administered Vaginally in the Treatment of Bacterial Vaginosis
Brief Title: Dose Ranging Study of SPL7013 Gel for Treatment of Bacterial Vaginosis (BV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Starpharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPL7013-013
Record Dates: First submitted 2010-08-30; First posted 2010-09-14 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Bacterial Vaginosis
Keywords: SPL7013; VivaGel; bacterial vaginosis; BV
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 0.5% SPL7013 Gel (Experimental)
  Interventions: Drug: 0.5% SPL7013 Gel
- 1.0% SPL7013 Gel (Experimental)
  Interventions: Drug: 1.0% SPL7013 Gel
- 3.0% SPL7013 Gel (Experimental)
  Interventions: Drug: 3.0% SPL7013 Gel
- Placebo Gel (Placebo Comparator)
  Interventions: Other: Placebo Gel

INTERVENTIONS:
Drug: 0.5% SPL7013 Gel — Vaginal gel
  Arms: 0.5% SPL7013 Gel
Drug: 1.0% SPL7013 Gel — Vaginal gel
  Arms: 1.0% SPL7013 Gel
Drug: 3.0% SPL7013 Gel — Vaginal gel
  Arms: 3.0% SPL7013 Gel
Other: Placebo Gel — Vaginal gel
  Arms: Placebo Gel

SUMMARY:
The purpose of this study is to determine the efficacy of SPL7013 Gel in the treatment of bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years with a diagnosis of BV according to Amsel's criteria and a Nugent score of ≥4
* Otherwise healthy

Exclusion Criteria:

* No active STIs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Macek, MD, Principal Investigator — contracted to Starpharma Pty Ltd
Locations (5):
- United States (5):
  - Precision Trials, Phoenix, Arizona
  - Downtown Women's Health Care, Denver, Colorado
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Bexar Clinical Trials, LLC, Irving, Texas
  - Tidewater Clinical Research Inc, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No relevant events.
Period: Overall Study
Arm/Group | 0.5% SPL7013 Gel | 1.0% SPL7013 Gel | 3.0% SPL7013 Gel | Placebo Gel
Started | 34 | 33 | 32 | 33
Completed | 32 | 29 | 27 | 29
Not Completed | 2 | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Population: modified intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5% SPL7013 Gel | 1.0% SPL7013 Gel | 3.0% SPL7013 Gel | Placebo Gel | Total
Number analyzed (Participants) | 30 | 27 | 26 | 28 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (7.68) | 30.0 (6.66) | 29.5 (7.24) | 30.6 (7.66) | 29.8 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 26 | 28 | 111
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 27 | 26 | 28 | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Women With Clinical Cure as a Measure of Efficacy
Description: Number of women with clinical cure as determined by absence of BV by the Amsel's criteria
Time Frame: Day 21-30
Population: The analysis population was the mITT. Patients with a missing assessment due to early withdrawal were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% SPL7013 Gel | 1.0% SPL7013 Gel | 3.0% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 30 | 26 | 25 | 26
Participants | 7 | 12 | 7 | 3
Statistical Analysis 1: Comparison: 1.0% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Women With Clinical Cure as a Measure of Efficacy
Description: Number of women with clinical cure as determined by absence of BV by the Amsel's criteria
Time Frame: Day 9-12
Population: The analysis population was the mITT. Patients with a missing assessment due to early withdrawal were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% SPL7013 Gel | 1.0% SPL7013 Gel | 3.0% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 29 | 27 | 24 | 27
Participants | 16 | 20 | 15 | 6
Statistical Analysis 1: Comparison: 1.0% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Number of Women With Nugent Cure as a Measure of Efficacy
Description: Number of women with Nugent cure, defined as a Nugent score 0-3 (normal flora), when a score of 7-10 (BV flora) was determined at Baseline.
Time Frame: Day 9-30
Population: The analysis population was the mITT. Patients with a missing assessment due to early withdrawal were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% SPL7013 Gel | 1.0% SPL7013 Gel | 3.0% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 29 | 26 | 25 | 27
Participants | 6 | 5 | 6 | 0
Statistical Analysis 1: Comparison: 1.0% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p = 0.025, Cochran-Mantel-Haenszel

4. Secondary Outcome: Patient Perceived Symptom Resolution as a Measure of Efficacy (Odor)
Description: Number of women with absence of patient-reported vaginal odor, as determined by responses in a symptom questionnaire as to whether or not they had vaginal odor.
Time Frame: Day 9-30
Population: The analysis population is the mITT.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% SPL7013 Gel | 1.0% SPL7013 Gel | 3.0% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 30 | 27 | 26 | 28
Participants | 20 | 21 | 21 | 8

5. Secondary Outcome: Incidence of Genital Adverse Events Potentially Related to Treatment
Description: Number of women who experience signs/symptoms of genital irritation potentially related to treatment, by solicited reporting of specific AEs as a measure of safety.
Time Frame: For the duration of the study (up to Visit Day 21-30)
Population: This outcome measure is adverse events, which are required to be reported separately under Adverse Events section.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% SPL7013 Gel | 1.0% SPL7013 Gel | 3.0% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 32 | 32 | 29 | 32
Participants | 6 | 5 | 6 | 6

ADVERSE EVENTS:
Arm/Group | 0.5% SPL7013 Gel | 1.0% SPL7013 Gel | 3.0% SPL7013 Gel | Placebo Gel
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 6/32 | 4/32 | 5/29 | 4/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5% SPL7013 Gel (N=32) | 1.0% SPL7013 Gel (N=32) | 3.0% SPL7013 Gel (N=29) | Placebo Gel (N=32)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 4 | 2 | 2 | 4
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 2 | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 1 | 3 | 1
Metrorrhagia (Reproductive system and breast disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a multicenter study, the PIs can only publish after the results of the trial have been published collectively.